CLINICAL TRIAL: NCT03082092
Title: Pre-operative Intravenous Steroid in Unilateral Primary Total Knee Replacement for Pain Relief and Recovery: A Double-Blind Randomized Controlled Trial
Brief Title: Pre-operative Intravenous Steroid in Total Knee Replacement for Pain Relief and Recovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Cheng Lok Yiu, Resident, Queen Elizabeth Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PISTKR
Record Dates: First submitted 2017-02-25; First posted 2017-03-17 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee; Pain; Recovery; Steroid; Replacement; Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Intervention Model Description: single-centre, double-blind, placebo-controlled randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients receiving elective unilateral primary total knee replacement in Queen Elizabeth Hospital during May 2017 to October 2017 will be assessed for eligibility according to the inclusion and exclusion criteria. 50 subjects will be recruited and randomized using computer into intervention group and placebo group by a nurse otherwise not involved in the trial. The randomization will be concealed in an opaque envelope.
  On the day of operation, a surgeon otherwise not involved in the trial will prepare the methylprednisolone and saline (placebo). The envelope will be opened by the list anesthetist. The operating surgeons, anesthetists, assessors (physiotherapists) and the patients were all blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone Group (Experimental): The intervention group will receive a single dose intravenous 125mg methylprednisolone diluted in 2.1ml of diluent on induction of total knee replacement.
  Interventions: Drug: Methylprednisolone Sodium Succinate
- Placebo Group (Placebo Comparator): The placebo group will receive a single dose intravenous 2.1ml of 0.9% IV saline, which is transparent and has no difference in appearance to methylprednisolone, on induction of total knee replacement
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Methylprednisolone Sodium Succinate — single intravenous dose of 125mg methylprednisolone diluted in 2.1ml of diluent given on induction of total knee replacement
  Arms: Methylprednisolone Group
Drug: Placebos — 0.9% intravenous saline (2.1ml) intravenously on induction of total knee replacement
  Arms: Placebo Group

SUMMARY:
Osteoarthritis of the knee is a common and important condition in our society. Despite various anesthetic methods and pain medications, pain after operation still remains as a challenge.

Steroids plays a role in decreasing the inflammatory reaction and stress response from surgery.

This study is to evaluate the use of an additional steroid injection, on top of usual pain killers and anesthesia, on the effect of pain control and recovery after total knee replacement.

50 subjects will be recruited, half of them will be randomized to receive a single dose of steroid injection before operation while the other half will receive a placebo. All the doctors, patients and physiotherapists are not aware of the allocation. Apart from the steroid or placebo injection, all the other treatment (eg: surgery, medications, rehabilitation protocol etc) will be the same. Doctors and physiotherapists will assess the subjects at 24, 30, 48 hours after surgery and upon discharge for their pain relief and recovery. Any complications will also be documented.

DETAILED DESCRIPTION:
Osteoarthritis of the knee is a common and important disease in the population. As a joint replacement centre, around 600 total knee replacements were performed in Queen Elizabeth Hospital and Buddhist Hospital per year. Despite multiple anesthetic methods and analgesics protocols, post-operative pain remains a significant problem.

Perioperative use of steroids has been shown to reduce postoperative nausea and vomiting. In both orthopaedic and non-orthopaedic operations, a single high dose of pre-operative steroid was also found to be effective in reducing early postoperative pain.

The hypothesis is that steroids help reduce post-operative inflammation and surgical stress response. Inflammatory markers such as IL-6 and C-reactive protein showed significant reduction after administration of perioperative steroids.

In a Denmark randomized-controlled trial published in 2010, the authors found that a single high-dose of methylprednisolone significantly reduce post-operative pain upto 48 hours in patients undergoing unilateral primary total knee replacement. Another randomized-controlled trial conducted in Korea in 2013 also showed significant pain control with less opioid consumption 6-24 hours after total knee replacement using dexamethasone. A group of United States researchers demonstrated that 3 doses of perioperative low dose hydrocortisone could also reduce post-bilateral total knee replacement pain at 24 hours with significant greater range of motion in a randomized-controlled trial published in 2012. However, there is no data on the effect of perioperative steroid use in Chinese population receiving total knee arthroplasty.

Upon induction, the intervention group will receive 125mg methylprednisolone diluted in 2.1ml of diluent intravenously. The placebo group will receive 2.1ml of 0.9% intravenous saline, which is transparent and has no difference in appearance to methylprednisolone.

All subjects will undergo total knee replacement using same implant (Zimmer NexGen LPS Flex) by same surgeons. All operations will be done under spinal anesthesia injecting 1.8-2.5ml 0.5% Bupivacaine into L3/4 or L4/5 disc space without fentanyl or other analgesics. Pre-operative, perioperative and postoperative analgesic regimen will be standardised.

Subjects will be assessed at 24, 30, 48 hours after surgery and upon discharge by physiotherapists. During each assessment, pain from operated knee will be assessed with 100mm visual analogue scale with patients performing different tasks, i.e.: at rest, maximal knee flexion, straight knee raise with 45 degree hip flexion, frame walking for 5m. Range of movement will also be documented in each assessment. Time to achieve independent frame walking and length of stay will be recorded in terms of days.

Analgesic consumption will be calculated with reference to the total amount of morphine administered through patient-controlled analgesia in the first 48 hours and the total dosage of rescue analgesia (DF118) required.

To assess the severity of inflammation, knee circumference (measured at the most superior border of patella in cm) will be measured before operation and 48 hours after operation. Biochemically, blood will be taken for C-reactive protein (CRP) in day 1 after surgery and compared with pre-operative CRP. Renal function and blood sugar will also be closely monitored to detect any hypokalaemia or hyperglycaemia. Subjects will also be asked to rate the sleep quality using a 100mm visual analogue scale (0 = worst sleep, 100 = best sleep).

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral total knee replacement for primary osteoarthritis of knee
* ASA (American Society of Anesthesiologists) grading 1 or 2

Exclusion Criteria:

* Rheumatoid arthritis or seronegative arthritis
* Allergy to any medications used in the standard protocol (Methylprednisolone, adrenaline, ropivacaine, ketorolac, bupivacaine, ketorolac, pepcidine, transamin, gabapentin, voltaren, panadol, DF118)
* Chronic opioid use
* Substance dependence
* Patients attending chronic pain clinic
* Psychiatric or neurological condition that may influence pain perception or reporting
* Chronic illness that preclude the use of the medications in the standard protocol
* Hepatitis B carrier or Elevated bilirubin or ALT
* Active peptic ulcer disease
* Uncontrolled diabetic patients with HbA1c >7% in recent 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Pain from operated knee using 100mm visual analogue scale | 24 hours after surgery
  during walking 5 metres with frame, using 100mm visual analogue scale

SECONDARY OUTCOMES:
Pain from operated knee (other than primary outcome) using 100mm visual analogue scale | 24 hours after surgery
  during rest, maximal knee flexion, straight knee raise with 45 degree hip flexion, using 100mm visual analogue scale
Pain from operated knee using 100mm visual analogue scale | 30 hours after surgery
  during rest, maximal knee flexion, straight knee raise with 45 degree hip flexion, walking 5 metres with frame, using 100mm visual analogue scale
Pain from operated knee using 100mm visual analogue scale | 48 hours after surgery
  during rest, maximal knee flexion, straight knee raise with 45 degree hip flexion, walking 5 metres with frame, using 100mm visual analogue scale
Pain from operated knee using 100mm visual analogue scale | upon discharge usually around post operative day 7
  during rest, maximal knee flexion, straight knee raise with 45 degree hip flexion, walking 5 metres with frame, using 100mm visual analogue scale
Range of movement from operated knee | 24, 30, 48 hours after surgery, upon discharge usually around post operative day 7
  Maximal knee flexion and maximal knee extension
Time to achieve independent frame walking | upon discharge usually around post operative day 7
  in terms of days
Length of stay | upon discharge usually around post operative day 7
  from day of admission to day of discharge, in terms of days
Patient-controlled analgesia consumption | 48 hours after surgery
  Total morphine use in patient-controlled analgesia
Rescue analgesics consumption | upon discharge usually around post operative day 7
  amount of rescue analgesics (DF118) needed
Knee circumference of the operated knee | 48 hours after surgery
  measured at most superior border of patella in cm
C-reactive Protein | day 1 after surgery
  blood taking for C-reactive protein
Sleep quality using 0-100 visual analogue scale | day 1 after surgery
  0-100 visual analogue scale, 0=worst sleep, 100= best sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng BLY, So EHK, Hui GKM, Yung BPK, Tsui ASK, Wang OKF, Poon MWY, Chan ACM, Wong SHS, Li W, Yip PSC. Pre-operative intravenous steroid improves pain and joint mobility after total knee arthroplasty in Chinese population: a double-blind randomized controlled trial. Eur J Orthop Surg Traumatol. 2019 Oct;29(7):1473-1479. doi: 10.1007/s00590-019-02469-5. Epub 2019 Jun 20. PMID 31222540